CLINICAL TRIAL: NCT05709548
Title: INDURG TRIAL: A Randomized Controlled Trial Using Indocyanine Green During Cholecystectomy in Acute Cholecystitis
Brief Title: Use of Indocyanine Green in Acute Cholecystitis
Acronym: INDURG
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Anna Muñoz - Campaña, Principal investigator, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INDURGTRIAL2022
Record Dates: First submitted 2023-01-12; First posted 2023-02-02 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Acute Cholecystitis; Bile Duct Injury
Keywords: Indocyanine green
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): patients who undergo urgent laparoscopic cholecystectomy according to the usual technique without the administration of indocyanine green
- intervention group (Active Comparator): Patients who undergo urgent laparoscopic cholecystectomy for acute cholecystitis with the administration of indocyanine green preoperatively.
  Interventions: Drug: Indocyanine green

INTERVENTIONS:
Drug: Indocyanine green — Subjects with a diagnosis of acute cholecystitis who undergo urgent laparoscopic cholecystectomy with the preoperative administration of indocyanine green (between 1-2 hours prior to surgery).
  Other Names: indocyanine green group
  Arms: intervention group

SUMMARY:
Laparoscopic cholecystectomy is one of the most common gastrointestinal surgeries. However, it can be technically complex in those patients diagnosed with acute cholecystitis who present severe inflammation or fibrosis, with bile duct injury being one of its main complications. The use of fluorescence cholangiography through the use of indocyanine green allows the identification of extrahepatic biliary structures, facilitating dissection and reducing the risk of bile duct lesions. Better visualization of the bile duct allows reducing the conversion rate to open surgery, as well as operating time.

The main objective is to assess a decrease in operating time in acute cholecystitis undergoing emergency surgery, to which indocyanine green is administered preoperatively.

Randomized, prospective, controlled, multicenter clinical trial of two groups of patients diagnosed with acute cholecystitis and requiring urgent cholecystectomy. The control group includes 220 patients who undergo urgent laparoscopic cholecystectomy according to the usual technique without the administration of indocyanine green, and the intervention group includes 220 patients who undergo urgent laparoscopic cholecystectomy for acute cholecystitis with the administration of indocyanine green preoperatively.

Study led by the Parc Taulí University Hospital in Sabadell.

DETAILED DESCRIPTION:
Prospective, controlled, randomized and multicenter clinical trial comparing conventional laparoscopic cholecystectomy versus laparoscopic cholecystectomy with preoperative indocyanine green administration in patients with an indication for urgent cholecystectomy due to acute cholecystitis (of any etiology), at the Parc Taulí University Hospital and at the Germans Trias i Pujol University Hospital.

Parallel group randomization (1:1) will be performed by opening sealed envelopes, with random assignment between the two groups (intervention and control). The same number of envelopes will be assigned to the study and control group, all of them sealed and placed at random.

A four-port laparoscopic cholecystectomy will be performed by a team of surgeons with extensive experience in emergency and/or hepatobiliopancreatic surgery, according to standard techniques and safety measures.

Randomization will be carried out at the time of the indication for surgery, after acceptance and signing of the informed consent once all the inclusion criteria are met.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication for urgent laparoscopic cholecystectomy due to acute cholecystitis regardless of its etiology.
* Age over 18 years.
* Patients who have read the study information sheet and signed the informed consent sheet.

Exclusion Criteria:

* Pregnant or breastfeeding patients.
* Grade IV renal failure or patients on dialysis
* Patients with previous hypersensitivity to indocyanine green
* Patients with allergy to iodinated contrast
* Patients with clinical hyperthyroidism, autonomic thyroid adenomas, and focal and diffuse autonomic abnormalities of the thyroid gland
* Contraindication to laparoscopic surgery.
* Suspicion of choledocholithiasis
* Pediatric patients under 18 years of age.
* Patients who refused to participate in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
operating time | from the beginning of the surgery to its end, up to 300 minutes
  time between the start of the surgical incision and the end of surgery

SECONDARY OUTCOMES:
admission days | length of hospital stay, from admission to discharge, up to 3 month
  days of hospital admission
intraoperative complications | during surgical time
  surgical injuries during surgery
postoperative morbidity | in the first 30 days after surgery
  complications evidenced in the postoperative period
visualization of biliary anatomy with indocyanine green | during surgical time
  Evidence the correct visualization of the biliary structures after the administration of indocyanine green

CONTACTS AND LOCATIONS:
Overall Officials: Anna Muñoz Campaña, PhD, Principal Investigator — Hospital Universitari Parc Taulí; Enrico Marrano, Principal Investigator — Germans Trias i Pujol Hospital
Locations (2):
- Spain (2):
  - Hospital Universitari Parc Tauli, Sabadell, Barcelona
  - Hospital de Vic, Vic, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pesce A, Piccolo G, Lecchi F, Fabbri N, Diana M, Feo CV. Fluorescent cholangiography: An up-to-date overview twelve years after the first clinical application. World J Gastroenterol. 2021 Sep 28;27(36):5989-6003. doi: 10.3748/wjg.v27.i36.5989. PMID 34629815
- [Background] Di Maggio F, Hossain N, De Zanna A, Husain D, Bonomo L. Near-Infrared Fluorescence Cholangiography can be a Useful Adjunct during Emergency Cholecystectomies. Surg Innov. 2022 Aug;29(4):526-531. doi: 10.1177/1553350620958562. Epub 2020 Sep 16. PMID 32936054
- [Background] Reeves JJ, Broderick RC, Lee AM, Blitzer RR, Waterman RS, Cheverie JN, Jacobsen GR, Sandler BJ, Bouvet M, Doucet J, Murphy JD, Horgan S. The price is right: Routine fluorescent cholangiography during laparoscopic cholecystectomy. Surgery. 2022 May;171(5):1168-1176. doi: 10.1016/j.surg.2021.09.027. Epub 2021 Dec 21. PMID 34952715
- [Background] Dip F, LoMenzo E, Sarotto L, Phillips E, Todeschini H, Nahmod M, Alle L, Schneider S, Kaja L, Boni L, Ferraina P, Carus T, Kokudo N, Ishizawa T, Walsh M, Simpfendorfer C, Mayank R, White K, Rosenthal RJ. Randomized Trial of Near-infrared Incisionless Fluorescent Cholangiography. Ann Surg. 2019 Dec;270(6):992-999. doi: 10.1097/SLA.0000000000003178. PMID 30614881
- [Background] Wang X, Teh CSC, Ishizawa T, Aoki T, Cavallucci D, Lee SY, Panganiban KM, Perini MV, Shah SR, Wang H, Xu Y, Suh KS, Kokudo N. Consensus Guidelines for the Use of Fluorescence Imaging in Hepatobiliary Surgery. Ann Surg. 2021 Jul 1;274(1):97-106. doi: 10.1097/SLA.0000000000004718. PMID 33351457
- [Background] Broderick RC, Lee AM, Cheverie JN, Zhao B, Blitzer RR, Patel RJ, Soltero S, Sandler BJ, Jacobsen GR, Doucet JJ, Horgan S. Fluorescent cholangiography significantly improves patient outcomes for laparoscopic cholecystectomy. Surg Endosc. 2021 Oct;35(10):5729-5739. doi: 10.1007/s00464-020-08045-x. Epub 2020 Oct 14. PMID 33052527
- [Background] van den Bos J, Schols RM, Luyer MD, van Dam RM, Vahrmeijer AL, Meijerink WJ, Gobardhan PD, van Dam GM, Bouvy ND, Stassen LP. Near-infrared fluorescence cholangiography assisted laparoscopic cholecystectomy versus conventional laparoscopic cholecystectomy (FALCON trial): study protocol for a multicentre randomised controlled trial. BMJ Open. 2016 Aug 26;6(8):e011668. doi: 10.1136/bmjopen-2016-011668. PMID 27566635
- [Background] Pavel MC, Boira MA, Bashir Y, Memba R, Llacer E, Estalella L, Julia E, Conlon KC, Jorba R. Near infrared indocyanine green fluorescent cholangiography versus intraoperative cholangiography to improve safety in laparoscopic cholecystectomy for gallstone disease-a systematic review protocol. Syst Rev. 2022 Mar 3;11(1):36. doi: 10.1186/s13643-022-01907-6. PMID 35241165